### TE 74/2022

### SHORT CHAIN FATTY ACIDS PROFILES IN AMYOTROPHIC LATERAL SCLEROSIS: LONGITUDINAL EFFECTS OF DISEASE AND MEDITERRANEAN DIET INTERVENTION

[IMPACT-ALS]

Project period 13/05/2022-12/05/2024

#### STUDY PROTOCOL

### SHORT CHAIN FATTY ACIDS PROFILES IN AMYOTROPHIC LATERAL SCLEROSIS: LONGITUDINAL EFFECTS OF DISEASE AND MEDITERRANEAN DIET INTERVENTION

## WP1 – Creation of the study design, informed consent for patients, definition of the study population and approval of the protocol

| WP1 | Objectives | Status |
|--------------|-------------------------------------|-----------|
| Deliverables | Establishment of the study protocol | Completed |
| | Ethics Committee approval | |
| | Informed consent form | Completed |

## WP2 - Determination of the reagents/materials needed at all stages of the research and initiation of procurement procedures

| WP 2 | Objectives | Status |
|---|---|---|
| Deliverables | Establishing the reagents and materials needed for the research stages (list of necessary materials and equipment, with technical specifications) Establishing the working protocol for neurophysiological exploration | Completed |
| | Commencement of procurement procedures, contact with suppliers | Completed |

# WP3 - Inclusion of patients in the study, initial visit (T0), clinical evaluation, neurophysiological evaluation, collection of biological samples and SCFA analysis (SCFAGGYC-PROF)

| WP 3 | Objectives | Status |
|------|------------|--------|

| Deliverables | Identification of patients with ALS (n=44) and healthy controls (similar age and gender; n=40) | Achieved |
|---|---|---|
| | Explaining the objectives of the study and signing the informed consent form | Completed |
| | Clinical and neurophysiological assessment of each ALS patient, with completion of each patient's medical record (including ALSFRS-R) | Completed |
| | Collection of serum samples | Completed |

# WP4 - Reassessment of ALS patients after 6 months (visit T1): clinical and neurophysiological evaluation, collection of biological samples and SCFA analysis, and introduction of the diet

| WP 4 | Objectives: Dissemination of research data | Status |
|--------------|-------------------------------------------------|-----------|
| | within the grant | |
| | Clinical and neurophysiological assessment of | Completed |
| | each ALS patient and application of the dietary | |
| | questionnaire | |
| Deliverables | Collection of serum samples | Completed |
| Denverables | Completion of the patient's medical file | Done |
| | Introduction of a dietary plan | Done |

## WP5 - Final reassessment of ALS patients (visit T2): clinical assessment, neurophysiological assessment, collection of biological samples and SCFA analysis

| WP 5 | Objectives | Status |
|---|---|---|
| Deliverables | Clinical and neurophysiological assessment of each ALS patient 6 months after introduction of the diet | Achieved |
| | Serum sample collection | Completed |
| | Completion of each patient's medical file | Completed |
| | Neurophysiological report | Done |

### WP6 - Serum analysis to identify serum SCFA levels

| WP 6 | Objectives: Analysis of stored plasma samples using specific analysis kits | Status |
|---|---|---|
| Deliverables | Plasma analysis sheets for the SCFAGGYC-PROF profile through the analysis of stored plasma samples Data entry into the database | Completed |

### WP 7 - Statistical analysis of collected data

| WP 7 | Objectives: Statistical analysis of clinical, paraclinical and electrophysiological data for each ALS patient compared to the control group | Status |
|---|---|---|
| Deliverables | Discovery of the SCFAGGYC-PROF profile in ALS patients at T0 compared to the control group; Discovery of the SCFAGGYC-PROF profile P-ALS in T0 and T1 evolution; Identification of changes in the dynamics of the SCFAGGYC-PROF profile in ALS patients comparing T0 with T2. | Achieved |